CLINICAL TRIAL: NCT01716208
Title: Phase II Trial of Ofatumumab and Fresh Frozen Plasma in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: Ofatumumab and Fresh Frozen Plasma in Patients With Chronic Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Tuscano (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Joseph Tuscano, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 333961; UCDCC#232 (Other Grant/Funding Number: UC Davis); OFT116066 (Other Grant/Funding Number: GlaxoSmithKline)
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Fresh Frozen Plasma; Complement; Monoclonal Antibody
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ofatumumab + Fresh Frozen Plasma (Experimental): Ofatumumab will be infused intravenously on day 1 (300 mg initial dose), followed one week later by 2000 mg weekly for 7 doses, followed 4 weeks later by 2000 mg every 4 weeks for 4 doses. Two units (approximately 200 or 250 ml) of FFP will be administered prior to ofatumumab(with the exception of the first dose). A unit of fresh frozen plasma is approximately 250ml (or half a pint).
  Interventions: Drug: Ofatumumab + Fresh Frozen Plasma

INTERVENTIONS:
Drug: Ofatumumab + Fresh Frozen Plasma
  Other Names: Azerra

SUMMARY:
It has been shown that many patients with lymphoma or chronic lymphocytic leukemia (CLL)have low levels of complement. Several drugs have been approved by the Food and Drug Administration (FDA) for use in this cancer. However, these drugs are often used as combination therapies which means two or more drugs are part of the treatment. Many people, especially elderly patients, cannot put up with the use of multiple drugs because of the side effects.

The main purpose of this study is to see if patients respond to therapy with human plasma (known as fresh frozen plasma or FFP) and ofatumumab. Another purpose of the study is to find out if this therapy will increase chances of getting rid of leukemia. This study will also look at the levels of complement in your blood. The levels of complement may allow better understanding of whether increasing the levels of complement by giving FFP may help control leukemia.

DETAILED DESCRIPTION:
The vast majority of patients with CLL are elderly and often they cannot tolerate standard multi-agent chemotherapeutic or biochemotherapeutic approaches. Based on this, less toxic and more effective treatment options are needed.

Ofatumumab has proven to be effective in patients with relapsed and/or refractory CLL. Previous studies have shown that ofatumumab is more effective than rituximab at activating complement and utilizing complement-dependent cytotoxicity (CDC).

This study will investigate treating relapsed/refractory CLL patients with FFP in combination with ofatumumab. The hypothesis is that patients with CLL have low complement levels and when they get treated with humanized antibodies like rituximab or ofatumumab these levels drop even further. Both these antibodies utilize complement to exert their cytotoxic effect, thus we hypothesize that by replacing complement levels with FFP we can enhance the efficacy of ofatumumab.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a pathological diagnosis of B-cell CLL.
* Patients must have received prior rituximab therapy and must have recovered from all non-hematologic toxicities. (Previous radiation is allowed as long as patients have recovered from all treatment related toxicities).
* Patients must meet the following laboratory values:

  * Hgb > 9.0 g/dl
  * Platelets > 50,000/mm3
  * Creatinine < 2.0 times the institutional upper limit of normal
  * SGOT/SGPT < 2.5 times the institutional upper limit of normal
  * Total Bilirubin <1. 5 times the institutional upper limit of normal
  * Alkaline phosphatase <2.5 times upper limit of normal (unless due to disease involvement of the liver or bone marrow)
* Patients must be at least 18 years of age.
* Patients must have a performance status of 0-2 by ECOG criteria.
* All patients must be informed of the investigational nature of this study and must sign and give written consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Subjects who have current active hepatic or biliary disease.
* Having received rituximab or rituximab-containing therapy within the prior 3 months.
* Treatment with any known therapeutic or experimental therapy within 4 weeks prior to enrollment, or currently participating in any other interventional clinical study.
* Other past or current malignancy.
* Prior treatment with anti-CD20 monoclonal antibody or alemtuzumab within 3 months prior to start of therapy.
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C.
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae.
* Known HIV positive.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure, and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient.
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg.
* Positive serology for hepatitis C (HC) defined as a positive test for HCAb, in which case reflexively perform a HC RIBA immunoblot assay on the same sample to confirm the result.
* Pregnant or lactating women.
* Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy.
* Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy.
* Receiving warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tuscano, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Comprehensive Cancer Center, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ofatumumab + Fresh Frozen Plasma: Ofatumumab will be infused intravenously on day 1 (300 mg initial dose), followed one week later by 2000 mg weekly for 7 doses, followed 4 weeks later by 2000 mg every 4 weeks for 4 doses. Two units (approximately 200 or 250 ml) of FFP will be administered prior to ofatumumab(with the exception of the first dose). A unit of fresh frozen plasma is approximately 250ml (or half a pint).
  Ofatumumab + Fresh Frozen Plasma
Period: Overall Study
Arm/Group | Ofatumumab + Fresh Frozen Plasma
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab + Fresh Frozen Plasma
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Response to Therapy
Description: Defined as complete, or partial response, and progression-free survival. Measured by National Cancer Institute - Working Group and International Workshop on Chronic Lymphocytic Leukemia
Time Frame: Up to 37 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab + Fresh Frozen Plasma
Number analyzed (Participants) | 12
Participants
  PR | 10
  CR | 2

2. Secondary Outcome: Number of Participants With Toxicities
Description: Toxicities will be graded according to the NCI CTCAE v4.0.
Time Frame: Up to two years
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab + Fresh Frozen Plasma
Number analyzed (Participants) | 12
Participants
  Blood bilirubin increased | 1
  Chills | 1
  Constipation | 1
  Cough | 1
  Creatinine increased | 2
  Dehydration | 1
  Dizziness | 2
  Dyspepsia | 1
  Dyspnea | 3
  Blepharitis | 1
  Fatigue | 5
  Flushing | 1
  Gastroesophageal reflux disease | 1
  Feverish | 1
  Generalized muscle weakness | 1
  Headache | 4
  Hiccups | 1
  Hyperkalemia | 1
  Hypertension | 2
  Hypocalcemia | 1
  hyponatremia | 1
  Infusion related reaction | 7
  Insomnia | 2
  Lung infection | 1
  Lymph node pain | 1
  Lymphocyte count increased | 2
  Nausea | 5
  Neutrophil count decreased | 4
  Palpitations | 1
  Paresthesia | 1
  peripheral sensory neuropathy | 1
  Platelet count decreased | 4
  Rash acneiform | 1
  Rash maculo-papular | 1
  Aspergillus Pneumonia | 1
  Sinus tachycardia | 1
  Sinusitis | 2
  Rash | 1
  Lesions on face, neck, scalp | 1
  Guttate Psoriasis (Exacerbation of Symptoms) | 1
  Skin infection, Eyelid | 4
  Upper respiratory infection | 1
  Wheezing | 1
  White blood cell decreased | 3

3. Secondary Outcome: Overall Survival
Description: Count of participants known to be alive up to two years from the time from start of treatment.
Time Frame: Up to two years
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab + Fresh Frozen Plasma
Number analyzed (Participants) | 12
Participants | 11

4. Secondary Outcome: Percent Reduction in Complement Levels (CH50)
Description: Complement CH50 is a blood test that helps us determine whether protein abnormalities and deficiencies in the complement system are responsible for any increase in autoimmune activity.
Time Frame: Up to two weeks
Measure: Mean (Full Range); unit: Percentage change
Arm/Group | Ofatumumab + Fresh Frozen Plasma
Number analyzed (Participants) | 12
Percentage change | 54 [20 to 100]

ADVERSE EVENTS:
Time Frame: Up to 2 years.
Description: Incidence of adverse events according to the Common Terminology Criteria for Adverse Events Version 4.0
Arm/Group | Ofatumumab + Fresh Frozen Plasma
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ofatumumab + Fresh Frozen Plasma (N=12)
Lung infection (Infections and infestations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab + Fresh Frozen Plasma (N=12)
Allergic reaction (Immune system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 3
Anxiety (Psychiatric disorders) | 1
Blood bilirubin increased (Investigations) | 1
Chills (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 2
Dyspspsia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Blepharitis (Eye disorders) | 1
Fatigue (General disorders) | 5
Flushing (Vascular disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Feverish (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 7
Insomnia (Psychiatric disorders) | 2
Lymph node pain (Blood and lymphatic system disorders) | 1
Lymphocyte count increased (Investigations) | 2
Nausea (Gastrointestinal disorders) | 5
Neutrophil count decreased (Investigations) | 4
Palpitations (Cardiac disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 4
Rash acneform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Aspergillus Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 4
Rash (Skin and subcutaneous tissue disorders) | 1
Guttate Psoriasis (Exacerbation of Symptoms) (Skin and subcutaneous tissue disorders) | 1
White blood cell decreased (Investigations) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT01716208/Prot_SAP_000.pdf